CLINICAL TRIAL: NCT00623922
Title: The Effect of Patient Education on Coping and Well Being in Patients With Arthritis.
Brief Title: Effect of Patient Education in Rheumatic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4.2007.2472; NSD 17975
Record Dates: First submitted 2008-02-12; First posted 2008-02-26 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Polyarthritis
Keywords: Patient education; Nurse consultation; Arthritis; Wellbeing; Coping; Health related quality of life
MeSH Terms: conditions — Arthritis | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patient education
  Interventions: Behavioral: Patient education with individual nurse consultations
- 2 (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Patient education with individual nurse consultations — 3 group meetings followed by 1-2 individual nurse consultations.
  Arms: 1

SUMMARY:
The purpose of this study is to explore the effect of patient education (PE) in patients with arthritis. PE has become a task that is dictated by law in Norway, and is increasingly used as an element in the treatment of patients with chronic complaints. Our hypothesis is that

- PE delivered as group education, followed by an individual nurse consultation increases the patients wellbeing an ability to cope with the disease.

DETAILED DESCRIPTION:
There has been a rather long tradition of PE for patients with arthritis. A recent systematic review found that PE had small short-term effects on disability, joint counts, patient global assessment, psychological status and depression, but this effect disappeared on the latest time of follow up (3-14 months). A recent large British study also failed to show an effect on pain, physical functioning, or contact with primary care after 12 months, but found a significant effect on anxiety and improved the participants' perceived self efficacy. This indicates that the present forms of interventions fails to show a long term effect. One possible reason for the lack of long term effect might be that these interventions are given to groups only. Patients seem to prefer one-to-one interaction regarding information about the disease and its treatment together with emotional aspects, while education in groups are preferred for physical training and relational topics.

ELIGIBILITY:
Inclusion Criteria:

* Polyarthritis
* 18-80 years
* native Norwegian speaking
* able to understand and participate in the PE program

Exclusion Criteria:

* Participated in a patient educational program the latest 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2008-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Self efficacy | Baseline, 4 and 12 months
Well being (Arizona Integrative Outcomes Scale) | Baseline, 4 and 12 months

SECONDARY OUTCOMES:
Arthritis Impact Measurement Scale 2 (affect, symptoms, social interaction, role) | Baseline, 4 and 12 months
The Hospital Anxiety and Depression Scale | Baseline, 4 and 12 months
Educational Needs Assessment Tools | Baseline, 4 and 12 months
Modified Health Assessment Questionnaire | Baseline, 4 and 12 months
DAS 28 score (Disease activity score) | Baseline, 4 and 12 months
Patient Activation Measurement (PAM) | Baseline, 4 and 12 months
Cost- benefit | Baseline, 4 and 12 months
Physical activity | Baseline, 4 and 12 months
Use of medications | Baseline, 4 and 12 months
fatigue (VAS scale) | Baseline, 4 and 12 months
Pain (VAS scale) | Baseline, 4 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, Principal Investigator — Norwegian University of Science and Technology; Kjersti Grønning, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology and St. Olavs Hospital HF, Trondheim, Trondheim, Norway

REFERENCES:
- [Background] Riemsma RP, Taal E, Kirwan JR, Rasker JJ. Systematic review of rheumatoid arthritis patient education. Arthritis Rheum. 2004 Dec 15;51(6):1045-59. doi: 10.1002/art.20823. No abstract available. PMID 15593105
- [Result] Gronning K, Skomsvoll JF, Rannestad T, Steinsbekk A. The effect of an educational programme consisting of group and individual arthritis education for patients with polyarthritis--a randomised controlled trial. Patient Educ Couns. 2012 Jul;88(1):113-20. doi: 10.1016/j.pec.2011.12.011. Epub 2012 Jan 23. PMID 22277625
- [Result] Gronning K, Rannestad T, Skomsvoll JF, Rygg LO, Steinsbekk A. Long-term effects of a nurse-led group and individual patient education programme for patients with chronic inflammatory polyarthritis - a randomised controlled trial. J Clin Nurs. 2014 Apr;23(7-8):1005-17. doi: 10.1111/jocn.12353. Epub 2013 Jul 22. PMID 23875718
- [Derived] Gronning K, Midttun L, Steinsbekk A. Patients' confidence in coping with arthritis after nurse-led education; a qualitative study. BMC Nurs. 2016 May 4;15:28. doi: 10.1186/s12912-016-0150-x. eCollection 2016. PMID 27147905